CLINICAL TRIAL: NCT04174300
Title: Molecular Response to Custom Manual Physiotherapy Treatment of Fibromyalgia & Chronic Fatigue Syndrome (CFS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Principal Investigator, María García Escudero, Professor, Fundación Universidad Católica de Valencia San Vicente Mártir
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCV/2018-2019/076
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Fibromyalgia (FM); Chronic Fatigue Syndrome (CFS)
Keywords: Manual Therapy; Physiotherapy; Fibromyalgia (FM); Chronic Fatigue Syndrome (CFS); RNAseq; microRNA; mechanomiR
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Masking Description: Outcome measures will be randomized and anonymized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manual Therapy (Experimental): 8 sessions of manual therapy (twice weekly) of 25 minutes including pressure maneuvers of about 4,5 N
  Interventions: Procedure: Manual Therapy

INTERVENTIONS:
Procedure: Manual Therapy — 8 sessions of manual therapy (twice weekly) of 25 minutes including pressure maneuvers of about 4,5 N
  Other Names: Physiotherapy treatment

SUMMARY:
Fibromyalgia (FM)and Chronic Fatigue Syndrome (CFS) are complex diseases often presenting overlapping symptomatology. Manual therapy (MT) protocols report benefits for pain treatment of FM, but the underlying mechanisms for patient improvement remain unknown.

The main goal of this study is to assess the molecular changes associating to mechanical and additional MT triggers, possibly involved in patient symptom improvement.

DETAILED DESCRIPTION:
Patients with Fibromyalgia as primary diagnosis assessed by the 1990 & 2010 ACR (American College of Rheumatology) criteria, presenting or not comorbid CFS, according to the Canadian and International CFS criteria, age 40-75 and BMI<35 (N=40), will be subjected to physiotherapy treatment consisting on 8 sessions of manual therapy (twice weekly) of 25 minutes including pressure maneuvers of about 4,5 N by a single operator (Collegiate Physiotherapist). Blood samples (10-20mls/participant) will be obtained before and after first treatment, and after fourth and last treatment to determine molecular blood changes associated to the physiotherapy protocol applied. PBMC (Peripheral Blood Molecular Cells) transcriptome before and after treatments (RNAseq) will be studied towards identifying treatment-associated differential expression, mechanomiR profiles included. Patient health status with treatment will be monitored by FIQ, MFI and SF-36 questionnaires, in addition to an anonymized satisfaction questionnaire to register potential undesired secondary effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FM with or without comorbid CFS
* Not receiving hormone therapy
* Not suffering from other diseases
* Without previous history of cancer
* Not actively participating in any pharmacological trial
* Not taking medication for at least 12 hours before blood draw
* Having signed informed consent

Exclusion Criteria:

- Any uncompliance with what is described as inclusion criteria

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Fatigue score | 8 weeks
  MFI, 1-5 scale (20 items), higher scores indicate higher degree of fatigue
Pain index | 8 weeks
  FIQ and Visual analogue scale (VAS) of pain, Scale 0-100, <39 mild, 39-58 moderate, ≥59 severe
Differential gene expression | 8 weeks
  RNAseq

SECONDARY OUTCOMES:
Quality of life score | 8 weeks
  SF-36, 0-100 Likert scale (36 items), lower scores indicate poorer quality of health
ANS (autonomic nervous system) dysfunction | 8 weeks
  Plantar pressure maps

OTHER OUTCOMES:
Subjective response to treatment | 8 weeks
  Custom-made questionnaire, -1 to +1 scale (ítems 1-5), scale 1-10 (item 6), 6 items total, higher scores indicate improvement of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Maria Garcia-Escudero, PhD, Principal Investigator — Catholic University of Valencia; Elisa Oltra, PhD, Study Chair — Catholic University of Valencia
Locations (1):
- Clinicas Universitarias UCV, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Espejo JA, Garcia-Escudero M, Oltra E. Unraveling the Molecular Determinants of Manual Therapy: An Approach to Integrative Therapeutics for the Treatment of Fibromyalgia and Chronic Fatigue Syndrome/Myalgic Encephalomyelitis. Int J Mol Sci. 2018 Sep 9;19(9):2673. doi: 10.3390/ijms19092673. PMID 30205597
- See also: UCV Physiotherapy Research Group — https://www.ucv.es/investigacion/grupos-de-investigacion/grupoclave/1431